CLINICAL TRIAL: NCT04718025
Title: Evaluation of Safety and Efficacy of Two Ticagrelor-based De-escalation Antiplatelet Strategies in Acute Coronary Syndrome: the Randomized, Multicenter, Double-blind ELECTRA RCT Study
Brief Title: Evaluation of Safety and Efficacy of Two Ticagrelor-based De-escalation Antiplatelet Strategies in Acute Coronary Syndrome
Acronym: ELECTRA-SIRIO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Jacek Kubica, Prof. dr hab., Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/ABM/01/00009
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: STEMI; NSTEMI; Unstable Angina
Keywords: ticagrelor; aspirin; acute coronary syndrome
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable; Acute Coronary Syndrome | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-dose ticagrelor with aspirin (LDTA) (Experimental): Patients with ACS in this arm will be subject to reduction of ticagrelor maintenance dose from 2x90mg to 2x60mg after the first month post-ACS, and will receive the following antiplatelet therapy:
  1. ticagrelor 2x90mg + aspirin 1x100mg during the first 30 days after ACS;
  2. ticagrelor 2x60mg + aspirin 1x100mg starting from day 31 until 12 months after ACS.
  Interventions: Drug: Ticagrelor 60mg; Drug: Aspirin
- Low-dose ticagrelor with placebo (LDTP) (Experimental): Patients with ACS in this arm will be subject to reduction of ticagrelor maintenance dose from 2x90mg to 2x60mg after the first month post-ACS, followed by discontinuation of aspirin after 3 months post-ACS, and will receive the following antiplatelet therapy:
  1. ticagrelor 2x90mg + aspirin 1x100mg during the first 30 days after ACS;
  2. ticagrelor 2x60mg + aspirin 1x100mg starting from day 31 until day 90 after ACS;
  3. ticagrelor 2x60mg + placebo starting from day 91 until 12 months after ACS.
  Interventions: Drug: Ticagrelor 60mg
- Standard-dose ticagrelor with aspirin (SDTA) (Active Comparator): Patients with ACS in this arm will receive standard dual antiplatelet therapy including ticagrelor 2x90mg + aspirin 1x100mg during the whole 12 months after ACS.
  Interventions: Drug: Ticagrelor 90mg; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor 90mg — Up to day 30 after ACS, all enrolled patients will receive standard-dose ticagrelor 2x90mg as a part of dual antiplatelet therapy. Participants in SDTA arm will continue treatment with ticagrelor 2x90mg until 12 months post-ACS, while patients in LDTA and LDTP will be switched to low-dose ticagrelor 2x60 mg starting on day 31.
  Other Names: Brilique
  Arms: Standard-dose ticagrelor with aspirin (SDTA)
Drug: Ticagrelor 60mg — Starting from day 31, LDTA and LDTP patients will receive low-dose ticagrelor 2x60mg until 12 months post-ACS.
  Other Names: Brilique
  Arms: Low-dose ticagrelor with aspirin (LDTA); Low-dose ticagrelor with placebo (LDTP)
Drug: Aspirin — Up to day 90 after ACS, all enrolled patients will receive aspirin 1x100mg as a part of dual antiplatelet therapy. Starting from day 91, LDTP patients will discontinue aspirin and proceed with low-dose ticagrelor monotherapy until 12 months post-ACS, while patients in LDTA and SDTA will continue aspirin 1x100 mg until 12 months post-ACS.
  Other Names: acetylsalicylic acid
  Arms: Low-dose ticagrelor with aspirin (LDTA); Standard-dose ticagrelor with aspirin (SDTA)

SUMMARY:
The ELECTRA-SIRIO 2 study is a randomized, multicenter, double-blind, investigator-initiated clinical trial aimed to evaluate safety and efficacy of two ticagrelor-based de-escalation antiplatelet strategies in patients with acute coronary syndrome (ACS). During the hospitalization due to ACS, participants will be randomized in a 1:1:1 ratio into one of three arms: low-dose ticagrelor with aspirin (LDTA), low-dose ticagrelor with placebo (LDTP), and standard-dose ticagrelor with aspirin (SDTA), the latter being the control arm. Up to day 30, all enrolled patients will receive standard-dose ticagrelor (2x90mg) + aspirin (1x100mg). Starting from day 31 LDTA and LDTP patients will receive low-dose ticagrelor (2x60mg) + aspirin (1x100mg), SDTA - continuation of previous treatment. Starting from day 91 LDTP patients will receive low-dose ticagrelor (2x60mg) + placebo, SDTA and LDTA - continuation of previous treatment. The aim of the study is to evaluate the influence of ticagrelor maintenance dose reduction from 2x90mg to 2x60mg with or without continuation of aspirin versus dual antiplatelet therapy with standard dose ticagrelor in reducing clinically relevant bleeding and maintaining anti-ischemic efficacy in ACS patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of STEMI or NSTEMI or unstable angina
* for patients with STEMI, the following three inclusion criteria will have to be met: 1) new ST-elevation at the J-point in two contiguous leads with the cut-point ≥1 mm in all leads other than leads V2-V3, where the following cut-points apply: ≥2mm in men ≥40 years; ≥2.5 mm in men <40 years, or ≥1.5 mm in women regardless of age; or a new left bundle-branch block 2) the intention to perform primary PCI 3) detection of a rise and/or fall of cardiac troponin values with at least one value above the 99th percentile upper reference limit
* for patients with NSTEMI or unstable angina, at least two of the following three criteria will have to be met:

  1. symptoms indicating myocardial ischaemia
  2. ST-segment changes on electrocardiography indicating myocardial ischaemia
  3. detection of a rise and/or fall of cardiac troponin values with at least one value above the 99th percentile upper reference limit in addition to at least one of the following:

  <!-- -->

  1. ≥60 years of age;
  2. previous MI or coronary artery by-pass grafting;
  3. ≥50% stenosis in ≥2 coronary arteries;
  4. previous ischaemic stroke or transient ischaemic attack;
  5. ≥50% carotid stenosis or cerebral revascularisation;
  6. diabetes mellitus;
  7. peripheral artery disease;
  8. chronic kidney disease with glomerular filtration rate <60 mL/min.

Exclusion Criteria:

* contraindications to ticagrelor or/and aspirin
* indications for oral anticoagulation therapy
* second or third grade atrio-ventricular block
* previous stent thrombosis on treatment with ticagrelor
* end stage kidney disease with glomerular filtration rate <15 mL/min or on haemodialysis
* administration of prasugrel during the index event
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
BARC type 2, 3 or 5 bleeding | 12 months after ACS
  The primary safety composite end point of this study is the first occurrence of type 2, 3 or 5 bleeding according to the BARC criteria, occurring during the first 12 months after ACS.
Death from any cause, nonfatal MI or nonfatal stroke. | 12 months after ACS
  The primary efficacy end point is the composite of death from any cause, first nonfatal MI, or first nonfatal stroke.

SECONDARY OUTCOMES:
Death from any cause, nonfatal MI, nonfatal stroke, BARC type 2, 3, or 5 bleeding. | 12 months after ACS
  The key secondary endpoint, net clinical effect, was defined as composite of death from any cause, nonfatal MI, or nonfatal stroke, and the first occurrence of BARC type 2, 3, or 5 bleeding.
BARC type 3 or 5 bleeding | 12 months after ACS
  Composite of the first occurrence of type 3 or 5 bleeding according to the BARC criteria.
TIMI major or minor bleeding | 12 months after ACS
  Composite of the first occurrence of major or minor bleeding according to the TIMI criteria.
GUSTO moderate, severe, or life-threatening bleeding | 12 months after ACS
  Composite of the first occurrence of moderate, severe, or life-threatening bleeding according to the GUSTO criteria.
ISTH major bleeding | 12 months after ACS
  The first occurrence of major bleeding according to the ISTH criteria.
Death from any cause | 12 months after ACS
  Death from any cause.
Death from cardiovascular causes | 12 months after ACS
  Death from cardiovascular causes.
Myocardial infarction | 12 months after ACS
  Occurrence of myocardial infarction.
Ischemic stroke | 12 months after ACS
  Occurrence of ischemic stroke.
Definite or probable stent thrombosis | 12 months after ACS
  Occurrence of definite or probable stent thrombosis
Dyspnea | 12 months after ACS
  Occurrence of dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, MD, PhD, Principal Investigator — Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Poland; Eliano Navarese, MD, PhD, Principal Investigator — Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Poland
Locations (1):
- Antoni Jurasz University Hospital No. 1, Bydgoszcz, Poland

REFERENCES:
- [Derived] Kubica J, Adamski P, Niezgoda P, Kubica A, Podhajski P, Baranska M, Uminska JM, Pietrzykowski L, Ostrowska M, Siller-Matula JM, Badariene J, Bartus S, Budaj A, Dobrzycki S, Fidor L, Gasior M, Gessek J, Gierlotka M, Gil R, Goracy J, Grzelakowski P, Hajdukiewicz T, Jaguszewski M, Janion M, Kasprzak J, Kern A, Klecha A, Kleinrok A, Kochman W, Krakowiak B, Legutko J, Lesiak M, Nosal M, Piotrowski G, Przybylski A, Roleder T, Skonieczny G, Sobieszek G, Tycinska A, Wojciechowski D, Wojakowski W, Wojcik J, Zielinska M, Zurakowski A, Specchia G, Gorog DA, Navarese EP. A new approach to ticagrelor-based de-escalation of antiplatelet therapy after acute coronary syndrome. A rationale for a randomized, double-blind, placebo-controlled, investigator-initiated, multicenter clinical study. Cardiol J. 2021;28(4):607-614. doi: 10.5603/CJ.a2021.0056. Epub 2021 Jun 7. PMID 34096012